CLINICAL TRIAL: NCT02753803
Title: A Randomized, Open-label, Multiple Dosing, Three-way Crossover Clinical Trial to Investigate the Pharmacokinetic/Pharmacodynamic Drug-drug Interaction of Evogliptin 5 mg and Pioglitazone 30 mg
Brief Title: Pharmacokinetic/Pharmacodynamic Drug-drug Interaction of Evogliptin 5 mg and Pioglitazone 30 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: DA1229_DIP_I
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A group (Experimental): Evogliptin Pioglitazone Evogliptin+Pioglitazone
  Interventions: Drug: Evogliptin, Pioglitazone, Evogliptin+Pioglitazone
- B group (Experimental): Pioglitazone Evogliptin Evogliptin+Pioglitazone
  Interventions: Drug: Pioglitazone, Evogliptin, Evogliptin+Pioglitazone
- C group (Experimental): Evogliptin Evogliptin+Pioglitazone Pioglitazone
  Interventions: Drug: Evogliptin, Evogliptin+Pioglitazone, Pioglitazone
- D group (Experimental): Pioglitazone Evogliptin+Pioglitazone Evogliptin
  Interventions: Drug: Pioglitazone, Evogliptin+Pioglitazone, Evogliptin
- E group (Experimental): Evogliptin+Pioglitazone Evogliptin Pioglitazone
  Interventions: Drug: Evogliptin+Pioglitazone, Evogliptin, Pioglitazone
- F group (Experimental): Evogliptin+Pioglitazone Pioglitazone Evogliptin
  Interventions: Drug: Evogliptin+Pioglitazone, Pioglitazone, Evogliptin

INTERVENTIONS:
Drug: Evogliptin, Pioglitazone, Evogliptin+Pioglitazone — Evogliptin : Evogliptin 5mg QD Pioglitazone : Pioglitazone 30mg QD Evogliptin+Pioglitazone : Evogliptin 5mg QD + Pioglitazone 30mg QD
  Other Names: Suganon; Actos
  Arms: A group
Drug: Pioglitazone, Evogliptin, Evogliptin+Pioglitazone — Pioglitazone : Pioglitazone 30mg QD Evogliptin : Evogliptin 5mg QD Evogliptin+Pioglitazone : Evogliptin 5mg QD + Pioglitazone 30mg QD
  Other Names: Suganon; Actos
  Arms: B group
Drug: Evogliptin, Evogliptin+Pioglitazone, Pioglitazone — Evogliptin : Evogliptin 5mg QD Evogliptin+Pioglitazone : Evogliptin 5mg QD + Pioglitazone 30mg QD Pioglitazone : Pioglitazone 30mg QD
  Other Names: Suganon; Actos
  Arms: C group
Drug: Pioglitazone, Evogliptin+Pioglitazone, Evogliptin — Pioglitazone : Pioglitazone 30mg QD Evogliptin+Pioglitazone : Evogliptin 5mg QD + Pioglitazone 30mg QD Evogliptin : Evogliptin 5mg QD
  Other Names: Suganon; Actos
  Arms: D group
Drug: Evogliptin+Pioglitazone, Evogliptin, Pioglitazone — Evogliptin+Pioglitazone : Evogliptin 5mg QD + Pioglitazone 30mg QD Evogliptin : Evogliptin 5mg QD Pioglitazone : Pioglitazone 30mg QD
  Other Names: Suganon; Actos
  Arms: E group
Drug: Evogliptin+Pioglitazone, Pioglitazone, Evogliptin — Evogliptin+Pioglitazone : Evogliptin 5mg QD + Pioglitazone 30mg QD Pioglitazone : Pioglitazone 30mg QD Evogliptin : Evogliptin 5mg QD
  Other Names: Suganon; Actos
  Arms: F group

SUMMARY:
A randomized, open-label, multiple dosing, three-way crossover clinical trial to investigate the pharmacokinetic/pharmacodynamic drug-drug interaction of evogliptin 5 mg and pioglitazone 30 mg after oral administration in healthy male subjects

DETAILED DESCRIPTION:
A randomized, open-label, multiple-dose, three-treatment, three-period, six-sequence, crossover study

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male Volunteers (Age: 19~45years)
* 55<Body Weight<90, 18<BMI<27
* FPG: 70-125 mg/dL

Exclusion Criteria:

* galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Clinically significant Medical History
* Allergy or Drug Hypersensitivity
* AST(SGOT), ALT(SGPT) > Upper Normal Range*1.5, eGFR<80 mL/min
* Drink during clinical trial period
* Smoking during clinical trial period
* Grapefruit/Caffeine intake during clinical trial period
* No Contraception

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
AUC | 1d~6d pre-dose, 15d~20d pre-dose, 29~34d pre-dose, 7d/21d/35d pre-dose and post-dose
  area under the concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Clinical Trials Center, Seoul National University Hospital
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided